CLINICAL TRIAL: NCT01436396
Title: Immunogenicity and Safety of Yellow Fever Vaccine (Stamaril®) Administered Concomitantly With Tetravalent Dengue Vaccine in Healthy Toddlers at 12-13 Months of Age in Colombia and Peru
Brief Title: Study of Yellow Fever Vaccine Administered With Tetravalent Dengue Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CYD29; U1111-1116-4913 (Other: WHO); 2014-001714-26 (EudraCT Number)
Record Dates: First submitted 2011-09-07; First posted 2011-09-19 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Hemorrhagic Fever; Yellow Fever
Keywords: Dengue; Dengue Hemorrhagic Fever; CYD Dengue Vaccines; Yellow Fever; Stamaril®; Flavivirus Infections
MeSH Terms: conditions — Dengue; Severe Dengue; Yellow Fever; Flavivirus Infections | interventions — Yellow Fever Vaccine; Vaccines; Measles-Mumps-Rubella Vaccine; Tetanus Toxoid; Haemophilus Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To ensure that objective safety data were obtained, the trial was designed using an observer-blind methodology since the products were visually different and may be recognized. For first trial vaccination (V01), the person who administered the injections knew which products were administered while either the participant or parent nor the Investigator in charge of safety evaluation knew which products were administered.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYD Dengue Vaccine Group (Experimental): Participants received the Stamaril® and the CYD dengue vaccine (Injection 1) at enrolment (Month [M] 0) at age 12 to 13 months; measles, mumps and rubella vaccine, pneumococcal conjugated vaccine, hepatitis A vaccine at M1 (age 13 to 14 months); CYD dengue vaccine (Injection 2) at M6 (age 18 to 19 months); diphtheria, tetanus, acellular pertussis, inactivated polio and Haemophilus influenza type b (DTaP-IPV/Hib) vaccine at M7 (age 19 to 20 months); and CYD dengue vaccine (Injection 3) at M12 (age 24 to 25 months); and hepatitis A vaccine at M13 (age 25 to 26 months).
  Interventions: Biological: Live, attenuated dengue serotype 1, 2, 3, and 4 virus; Biological: Yellow fever vaccine; Biological: Measles, mumps, and rubella (MMR) vaccine; Biological: Pneumococcal Conjugated Vaccine; Biological: Hepatitis A Pediatric Vaccine; Biological: Diphtheria, tetanus, pertussis, polio, and Haemophilus influenzae vaccine
- Placebo Group (Experimental): Participants received the Stamaril® vaccine and placebo matched to CYD vaccine (Injection 1) at enrolment (M0) (age 12 to 13 months); measles, mumps, and rubella vaccine, pneumococcal conjugate vaccine and hepatitis A vaccine at M1 (age 13 to 14 months); CYD dengue vaccine (Injection 2) at M6 (age 18 to 19 months); DTaP IPV/Hib vaccine at M7 (age19 to 20 months); and CYD dengue vaccine (Injection 3) at M12 (age 24 to 25 months); and hepatitis A vaccine at M13 (age 25 to 26 months).
  Interventions: Biological: Live, attenuated dengue serotype 1, 2, 3, and 4 virus; Biological: Yellow Fever Vaccine; Biological: Placebo (NaCl); Biological: Measles, mumps, and rubella vaccine; Biological: Pneumococcal Conjugated Vaccine; Biological: Diphtheria, tetanus, pertussis, polio, and Haemophilus influenzae vaccine; Biological: Hepatitis A Pediatric Vaccine

INTERVENTIONS:
Biological: Live, attenuated dengue serotype 1, 2, 3, and 4 virus — 0.5 mL, subcutaneous at age 12, 18, and 24 months
  Other Names: CYD Dengue Vaccine
  Arms: CYD Dengue Vaccine Group
Biological: Yellow fever vaccine — 0.5 mL subcutaneous in the deltoid at age 12 to 13 months.
  Other Names: Stamaril®
  Arms: CYD Dengue Vaccine Group
Biological: Measles, mumps, and rubella (MMR) vaccine — 0.5 mL, subcutaneous at age 12 to 13 months.
  Other Names: MMR vaccine
  Arms: CYD Dengue Vaccine Group
Biological: Pneumococcal Conjugated Vaccine — 0.5 mL, intramuscular at age 13 to 14 months
  Arms: CYD Dengue Vaccine Group
Biological: Hepatitis A Pediatric Vaccine — 0.5 mL, intramuscular at age 13 to 14 months and 25 to 26 months
  Arms: CYD Dengue Vaccine Group
Biological: Diphtheria, tetanus, pertussis, polio, and Haemophilus influenzae vaccine — 0.5 mL, intramuscular at age 19 to 20 months
  Other Names: DTaP IPV//Hib Vaccine
  Arms: CYD Dengue Vaccine Group
Biological: Live, attenuated dengue serotype 1, 2, 3, and 4 virus — 0.5 mL, subcutaneous at age 18 to 19 and 24 to 25 months
  Other Names: CYD dengue vaccine
  Arms: Placebo Group
Biological: Yellow Fever Vaccine — 0.5 mL, subcutaneous at age 12 to 13 months
  Other Names: Stamaril®
  Arms: Placebo Group
Biological: Placebo (NaCl) — 0.5 mL, subcutaneous at age 12 to 13 months
  Other Names: NaCl 0.9%
  Arms: Placebo Group
Biological: Measles, mumps, and rubella vaccine — 0.5 mL, subcutaneous at age 13 to 14 months
  Other Names: MMR vaccine
  Arms: Placebo Group
Biological: Pneumococcal Conjugated Vaccine — 0.5 mL, intramuscular at age 13 to 14 months
  Arms: Placebo Group
Biological: Diphtheria, tetanus, pertussis, polio, and Haemophilus influenzae vaccine — 0.5 mL, intramuscular at age 19 to 20 months
  Other Names: DTaP IPV//Hib Vaccine
  Arms: Placebo Group
Biological: Hepatitis A Pediatric Vaccine — 0.5 mL, intramuscular at age 13 to 14 months and 25 to 26 months
  Arms: Placebo Group

SUMMARY:
The study was designed to evaluate whether the first CYD dengue vaccination can be administered concomitantly with Stamaril® yellow fever vaccine during the same day and visit, but at 2 different sites of administration.

Primary Objective:

* To demonstrate the non-inferiority of the immune response against Yellow Fever (YF) in flavivirus (FV) non-immune subjects at baseline receiving one dose of Stamaril vaccine administered concomitantly with the first dose of CYD dengue vaccine compared to participants receiving one dose of Stamaril vaccine concomitantly with placebo.

Secondary Objectives:

* To assess the non-inferiority of YF immune response 28 days post-Stamaril vaccination based on seroconversion rates regardless of the FV status of participants at baseline.
* To describe the YF immune response 28 days post-Stamaril vaccination in both groups.
* To describe the antibody (Ab) response to each dengue virus serotype 28 days post CYD dengue vaccine (Visit [V] 05 and V07), following CYD dengue vaccine Dose 1 and Dose 2 from Group 2 versus following CYD dengue vaccine Dose 2 and Dose 3 for Group 1 (effect of YF vaccination).
* To describe the safety of Stamaril vaccine administered concomitantly with the first dose of CYD dengue vaccine, or Stamaril administered concomitantly with placebo.
* To describe the safety of CYD dengue vaccine after the first dose of CYD dengue vaccine administered concomitantly with Stamaril vaccine or CYD vaccine administered alone.
* To describe the safety of the CYD dengue vaccine in all participants after each dose.

DETAILED DESCRIPTION:
All participants received a total of 9 injections during the study. Vaccine immunogenicity assessments for dengue neutralizing antibodies was performed in a randomized subset of participants. All participants were followed-up for safety during the study and for 6 months after the last CYD dengue vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 13 months on the day of inclusion.
* Born at full term of pregnancy (>=37 weeks) and with a birth weight >=2.5 kg as reported by the parent/legally acceptable representative.
* Participant in good health, based on medical history and physical examination.
* Participant had completed his/her vaccination schedule according to the official immunization calendar of Colombia and/or Peru, respectively.
* Informed consent form had been signed and dated by the parent(s) or other legally acceptable representative (and by 2 independent witnesses if required by local regulations).
* Participant and parent/legally acceptable representative/tutor able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Planned receipt of any vaccine in the 4 weeks following first trial vaccination.
* Previous vaccination against YF, hepatitis A, or measles, mumps and rubella.
* Receipt of blood or blood-derived products in the past 3 months which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 weeks or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Personal known seropositivity for human immunodeficiency virus (HIV) as reported by the parent/legally acceptable representative.
* History of previous maternal vaccination against YF as reported by the parent/legally acceptable representative.
* Personal history of YF or dengue infection/disease as reported by the parent/legally acceptable representative.
* Known systemic hypersensitivity to any of the vaccine components of the vaccines that were used in the trial, or history of a life-threatening reaction to the vaccines used in the trial or to vaccines containing any of the same substances.
* History of contraindication to receipt of vaccines containing components of Stamaril® (yellow fever vaccine), measles, mumps and rubella vaccine, hepatitis A vaccine, pneumococcal conjugated vaccine or of diphtheria (D) toxoid, tetanus (T) toxoid, pertussis toxoid (PT), filamentous hemagglutinin (FHA), polyribosylribitol phosphate (PRP) and polio or other diphtheria, tetanus and pertussis vaccine (e.g., DTwP).
* Thrombocytopenia, as reported by the parent/legally acceptable representative.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular (IM) vaccination.
* History of central nervous system disorder or disease, including seizures.
* Personal history of thymic pathology (e.g., thymoma), and/or thymectomy.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Identified as a child (adopted or natural) of the Investigator or of employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center.

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 792 (Actual)
Dates: Start 2011-09-07 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Cali, Colombia
- Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 07 September 2011 to 08 March 2012 at 2 clinical sites (1 in Colombia and 1 in Peru).
Pre-assignment Details: A total of 792 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized; 787 participants were vaccinated.
Groups:
- CYD Dengue Vaccine Group: Participants received the Stamaril® and the CYD dengue vaccine (Injection [Inj.] 1) at enrolment (M0) at age 12 to 13 months; measles, mumps and rubella vaccine, pneumococcal conjugated vaccine, hepatitis A vaccine at M1 (age 13 to 14 months); CYD dengue vaccine (Injection 2) at M6 (age 18 to 19 months); diphtheria, tetanus, acellular pertussis, inactivated polio and Haemophilus influenza type b (DTaP IPV/Hib) vaccine at M7 (age 19 to 20 months); and CYD dengue vaccine (Injection 3) at M12 (age 24 to 25 months); and hepatitis A vaccine at M13 (age 25 to 26 months).
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 396 | 396
Vaccinated | 394 | 393
Completed | 364 | 354
Not Completed | 32 | 42
Not completed — Protocol Violation | 7 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 19 | 29
Not completed — Serious adverse event | 2 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Safety Analysis Set which included all participants who had received at least 1 dose of CYD dengue vaccine, stamaril® vaccine or placebo.
Groups:
- CYD Dengue Vaccine Group: Participants received the Stamaril® and the CYD dengue vaccine (Injection 1) at enrolment (M0) at age 12 to 13 months; measles, mumps and rubella vaccine, pneumococcal conjugated vaccine, hepatitis A vaccine at M1 (age 13 to 14 months); CYD dengue vaccine (Injection 2) at M6 (age 18 to 19 months); diphtheria, tetanus, acellular pertussis, inactivated polio and Haemophilus influenza type b (DTaP IPV/Hib) vaccine at M7 (age 19 to 20 months); and CYD dengue vaccine (Injection 3) at M12 (age 24 to 25 months); and hepatitis A vaccine at M13 (age 25 to 26 months).
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 394 | 393 | 787
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 394 | 393 | 787
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.2 (0.25) | 12.2 (0.25) | 12.2 (0.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 203 | 401
  Male | 196 | 190 | 386

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Flavi Virus (FV) Non-immune Participants With Seroconversion Against YF Antigen After Vaccination With Yellow Fever (YF) Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Neutralizing antibodies against YF were assessed using a YF virus plaque reduction neutralization test (YF PRNT50) assay. Seroconversion was defined as YF antibodies >=10 (1/dilution [dil]) in flavivirus non-immune participants (defined as those with YF antibodies <10 [1/dil] for all serotypes (Serotype 1, 2, 3 and 4) with parental dengue virus strains and for YF virus).
Time Frame: 28 days Post-Injection 1
Population: Analysis was performed on Per-Protocol analysis set which included all participants who had no protocol deviations. Per-Protocol analysis set was defined for the Stamaril® vaccine immune response.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 296 | 299
Percentage of participants | 100.0 | 99.7
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; Non-inferiority of YF seroconversion rate was assessed 28 days post-Stamaril®/CYD dengue vaccine (CYD Dengue Vaccine Group) or post-Stamaril®/placebo (Placebo Group); Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 95% Confidence Interval (CI) was greater than -10. The difference in percentage of seroconversion rates between group 1 and 2 was based on the Wilson score (without continuity adjustment) 95% two-sided CI; Difference in percentage = 0.334, 95% CI 2-sided [-0.976 to 1.87]

2. Secondary Outcome: Percentage of All Participants With Seroconversion Against YF Antigen After Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Neutralizing antibodies against YF were assessed using a YF virus plaque reduction neutralization test (YF PRNT50) assay. Seroconversion was defined as YF antibodies >= 10 (1/dil) in participants YF-seronegative at baseline or 4-fold increase from pre- to post-YF antibody titers in participants YF-seropositive at baseline.
Time Frame: 28 days Post-Injection 1
Population: Analysis performed on Full analysis set included participants who received at least co-administration of Stamaril® vaccine with either 1st dose of CYD dengue vaccine or placebo, had blood sample post-Stamaril® vaccination drawn and a valid test result. Here, 'overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 378 | 376
Percentage of participants | 98.7 | 99.7
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 95% CI is greater than -10. The difference in percentage of seroconversion rates between group 1 and 2 was based on the Wilson score (without continuity adjustment) 95% two-sided CI; Difference in percentage = -1.06, 95% CI 2-sided [-2.81 to 0.383]

3. Secondary Outcome: Geometric Mean Titers (GMTs) of YF Antibodies in All Participants Following Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: GMTs against YF were assessed using a YF virus plaque reduction neutralization test (YF PRNT50) assay.
Time Frame: Pre-Injection 1 and 28-days Post-Injection 1
Population: Analysis was performed on Full analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 381 | 377
Titers (1/dilution)
  Pre-Injection 1: number analyzed (Participants) | 378 | 376
  Pre-Injection 1 | 5.64 [5.41 to 5.89] | 5.67 [5.42 to 5.93]
  Post-Injection 1 | 369 [322 to 423] | 423 [375 to 478]

4. Secondary Outcome: Geometric Mean Titer Ratios (GMTRs) of YF Antibodies in All Participants Following Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: GMTs ratios against YF were assessed using a YF virus plaque reduction neutralization test (YF PRNT50) assay.
Time Frame: Pre-Injection 1 and 28- days Post-Injection 1
Population: Analysis was performed on Full analysis set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure."
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 378 | 376
Ratio | 35.1 [30.5 to 40.4] | 39.8 [35.3 to 45.0]

5. Secondary Outcome: Percentage of All Participants With YF Antibody Titers of >=10 (1/Dil) Before and After Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Neutralizing antibodies against YF were assessed using a YF virus plaque reduction neutralization test (YF PRNT50) assay. Seroconversion was defined as YF antibodies >=10 (1/dil) regardless of the flavivirus status of participants at baseline.
Time Frame: Pre-Injection 1 and 28-days Post-Injection 1
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 381 | 377
Percentage of participants
  Pre-Injection 1: number analyzed (Participants) | 378 | 376
  Pre-Injection 1 | 9.0 | 9.0
  Post-Injection 1 | 99.5 | 99.7

6. Secondary Outcome: GMTs of Dengue Virus Antibodies Following Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: GMTs against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue plaque reduction neutralization test (PRNT) assay.
Time Frame: Pre-Injection 1 and 28-days Post-Injections 2 and 3
Population: Analysis performed on Full analysis set for dengue immunogenicity which included participants who received at least 1dose of CYD dengue vaccine/placebo, had at least 1 blood sample withdrawn and valid post vaccination test results for at least 1 dengue serotype. Here,'number analyzed' =participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 113
Titers (1/dilution)
  Serotype 1; Pre-Injection 1: number analyzed (Participants) | 109 | 110
  Serotype 1; Pre-Injection 1 | 5.08 [4.92 to 5.25] | 5.00 [5.00 to 5.00]
  Serotype 1; Post-Injection 2 | 47.3 [38.9 to 57.5] | 11.8 [9.82 to 14.1]
  Serotype 1; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 1; Post-Injection 3 | 89.0 [76.4 to 104] | 61.3 [52.5 to 71.5]
  Serotype 2; Pre-Injection 1: number analyzed (Participants) | 109 | 107
  Serotype 2; Pre-Injection 1 | 5.10 [4.96 to 5.23] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-Injection 2 | 95.5 [78.0 to 117] | 41.1 [33.2 to 51.0]
  Serotype 2; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 2; Post-Injection 3 | 173 [142 to 211] | 150 [127 to 177]
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 106 | 109
  Serotype 3; Pre-Injection 1 | 5.05 [4.95 to 5.16] | 5.18 [5.00 to 5.37]
  Serotype 3; Post-Injection 2 | 118 [101 to 137] | 43.4 [36.0 to 52.3]
  Serotype 3; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 3; Post-Injection 3 | 181 [158 to 207] | 155 [136 to 176]
  Serotype 4; Pre-Injection 1: number analyzed (Participants) | 110 | 112
  Serotype 4; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.05 [4.96 to 5.14]
  Serotype 4; Post-Injection 2 | 68.1 [54.6 to 84.9] | 29.8 [22.1 to 40.2]
  Serotype 4; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 4; Post-Injection 3 | 74.0 [61.3 to 89.4] | 74.6 [62.5 to 89.1]

7. Secondary Outcome: GMTRs of Dengue Virus Antibodies Following Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: GMTRs against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue PRNT assay.
Time Frame: Pre-Injection 1 and 28-days Post-Injections 2 and 3
Population: Analysis was performed on Full analysis set for dengue immunogenicity. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratios
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 113
Titer ratios
  Serotype 1; Post-Inj.2/Pre-Inj. 1: number analyzed (Participants) | 109 | 110
  Serotype 1; Post-Inj.2/Pre-Inj. 1 | 4.78 [3.91 to 5.84] | 1.15 [0.973 to 1.37]
  Serotype 1; Post-Inj.3/Pre-Inj. 1: number analyzed (Participants) | 107 | 104
  Serotype 1; Post-Inj.3/Pre-Inj. 1 | 8.82 [7.55 to 10.3] | 6.14 [5.26 to 7.18]
  Serotype 2; Post-Inj.2/Pre-Inj. 1: number analyzed (Participants) | 109 | 107
  Serotype 2; Post-Inj.2/Pre-Inj. 1 | 9.55 [7.75 to 11.8] | 3.86 [3.15 to 4.72]
  Serotype 2; Post-Inj.3/Pre-Inj. 1: number analyzed (Participants) | 107 | 102
  Serotype 2; Post-Inj.3/Pre-Inj. 1 | 16.7 [13.7 to 20.4] | 15.2 [12.8 to 18.1]
  Serotype 3; Post-Inj.2/Pre-Inj. 1: number analyzed (Participants) | 106 | 109
  Serotype 3; Post-Inj.2/Pre-Inj. 1 | 11.6 [9.98 to 13.5] | 4.16 [3.46 to 5.00]
  Serotype 3; Post-Inj.3/Pre-Inj. 1: number analyzed (Participants) | 104 | 104
  Serotype 3; Post-Inj.3/Pre-Inj. 1 | 18.0 [15.6 to 20.8] | 15.4 [13.5 to 17.6]
  Serotype 4; Post-Inj.2/Pre-Inj. 1: number analyzed (Participants) | 110 | 112
  Serotype 4; Post-Inj.2/Pre-Inj. 1 | 6.82 [5.44 to 8.55] | 2.89 [2.15 to 3.89]
  Serotype 4; Post-Inj.3/Pre-Inj. 1: number analyzed (Participants) | 108 | 106
  Serotype 4; Post-Inj.3/Pre-Inj. 1 | 7.26 [6.02 to 8.77] | 7.44 [6.24 to 8.88]

8. Secondary Outcome: Percentage of Participants With Antibody Titer >= 10 (1/Dil) Against Each Serotype With Parental Dengue Virus Strains After Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Neutralizing antibodies against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue PRNT assay. Seroconversion was defined as antibody titers >= 10 (1/dil) against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains.
Time Frame: Pre-Injection 1 and 28-days Post-Injections 2 and 3
Population: Analysis was performed Full analysis set for dengue immunogenicity. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 113
Percentage of participants
  Serotype 1; Pre-Injection 1: number analyzed (Participants) | 109 | 110
  Serotype 1; Pre-Injection 1 | 0.9 | 0.0
  Serotype 1; Post-Injection 2 | 92.0 | 51.3
  Serotype 1; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 1; Post-Injection 3 | 100.0 | 97.2
  Serotype 2; Pre-Injection 1: number analyzed (Participants) | 109 | 107
  Serotype 2; Pre-Injection 1 | 1.8 | 0.0
  Serotype 2; Post-Injection 2 | 97.3 | 86.7
  Serotype 2; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 2; Post-Injection 3 | 100.0 | 100.0
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 106 | 109
  Serotype 3; Pre-Injection 1 | 0.9 | 3.7
  Serotype 3; Post-Injection 2 | 100.0 | 90.3
  Serotype 3; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 3; Post-Injection 3 | 100.0 | 100.0
  Serotype 4; Pre-Injection 1: number analyzed (Participants) | 110 | 112
  Serotype 4; Pre-Injection 1 | 0.0 | 0.9
  Serotype 4; Post-Injection 2 | 91.2 | 68.1
  Serotype 4; Post-Injection 3: number analyzed (Participants) | 110 | 106
  Serotype 4; Post-Injection 3 | 97.3 | 98.1

9. Secondary Outcome: Percentage of Participants With Antibody Titer >= 10 (1/Dil) Against at Least 1, 2, 3, or 4 Serotypes With Parental Dengue Virus Strains After YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Neutralizing antibodies against at least 1, 2, 3, or 4 serotypes (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue PRNT assay.
Time Frame: Pre-Injection 1 and 28 days Post-Injections 2 and 3
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 113
Percentage of participants
  At least 1 serotype; Pre-Injection 1: number analyzed (Participants) | 111 | 112
  At least 1 serotype; Pre-Injection 1 | 3.6 | 4.5
  At least 1 serotype; Post-Injection 2 | 100.0 | 93.8
  At least 1 serotype; Post-Injection 3: number analyzed (Participants) | 110 | 106
  At least 1 serotype; Post-Injection 3 | 100.0 | 100.0
  At least 2 serotypes; Pre-Injection 1: number analyzed (Participants) | 111 | 112
  At least 2 serotypes; Pre-Injection 1 | 0.0 | 0.0
  At least 2 serotypes; Post-Injection 2 | 100.0 | 87.6
  At least 2 serotypes; Post-Injection 3: number analyzed (Participants) | 110 | 106
  At least 2 serotypes; Post-Injection 3 | 100.0 | 100.0
  At least 3 serotypes; Pre-Injection 1: number analyzed (Participants) | 111 | 112
  At least 3 serotypes; Pre-Injection 1 | 0.0 | 0.0
  At least 3 serotypes; Post-Injection 2 | 94.7 | 73.5
  At least 3 serotypes; Post-Injection 3: number analyzed (Participants) | 110 | 106
  At least 3 serotypes; Post-Injection 3 | 100.0 | 98.1
  All 4 serotypes; Pre-Injection 1: number analyzed (Participants) | 111 | 112
  All 4 serotypes; Pre-Injection 1 | 0.0 | 0.0
  All 4 serotypes; Post-Injection 2 | 85.8 | 41.6
  All 4 serotypes; Post-Injection 3: number analyzed (Participants) | 110 | 106
  All 4 serotypes; Post-Injection 3 | 97.3 | 97.2

10. Secondary Outcome: GMTs of Dengue Virus Antibodies of FV Immune Participants Following Vaccination With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: GMTs against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue PRNT assay. FV immune participants at baseline were defined as those participants with >= 10 (1/dil) for at least 1 serotype with the parental dengue virus strain or for YF virus.
Time Frame: Pre-Injection 1 and 28 days Post-Injections 2 and 3
Population: Analysis was performed on Full analysis set for dengue immunogenicity. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 10 | 14
Titers (1/dilution)
  Serotype 1; Pre-Injection 1: number analyzed (Participants) | 10 | 13
  Serotype 1; Pre-Injection 1 | 5.96 [4.01 to 8.87] | 5.00 [5.00 to 5.00]
  Serotype 1; Post-Injection 2 | 52.5 [25.0 to 110] | 17.0 [7.63 to 38.0]
  Serotype 1; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 1; Post-Injection 3 | 81.7 [47.3 to 141] | 59.5 [44.6 to 79.5]
  Serotype 2; Pre-Injection 1: number analyzed (Participants) | 10 | 12
  Serotype 2; Pre-Injection 1 | 6.14 [4.50 to 8.38] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-Injection 2 | 72.4 [47.4 to 111] | 74.3 [27.6 to 200]
  Serotype 2; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 2; Post-Injection 3 | 110 [75.5 to 160] | 133 [95.7 to 186]
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 8 | 13
  Serotype 3; Pre-Injection 1 | 5.74 [4.15 to 7.94] | 6.75 [5.05 to 9.03]
  Serotype 3; Post-Injection 2 | 102 [54.8 to 189] | 95.8 [61.3 to 150]
  Serotype 3; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 3; Post-Injection 3 | 143 [89.7 to 227] | 126 [91.7 to 173]
  Serotype 4; Pre-Injection 1: number analyzed (Participants) | 10 | 13
  Serotype 4; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.41 [4.55 to 6.43]
  Serotype 4; Post-Injection 2 | 87.1 [36 to 210] | 109 [44.7 to 265]
  Serotype 4; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 4; Post-Injection 3 | 77.1 [24.0 to 248] | 74.3 [40.9 to 135]

11. Secondary Outcome: GMTs of Dengue Virus Antibodies of FV-Non Immune (Naïve) Participants Following Vaccination With YF Vaccine Non Immune (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: GMTs against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue PRNT assay. FV-non-immune participants at baseline were defined as those participants with <10 (1/dil) for all serotypes (Serotype 1, 2, 3 and 4) with parental dengue virus strains and for YF virus.
Time Frame: Pre-Injection 1 and 28 days Post-Injections 2 and 3
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 94 | 90
Titers (1/dilution)
  Serotype 1; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 1; Post-Injection 2 | 45.9 [37.0 to 57.0] | 11.4 [9.42 to 13.7]
  Serotype 1; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 1; Post-Injection 3 | 86.6 [73.0 to 103] | 61.8 [51.5 to 74.3]
  Serotype 2; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-Injection 2 | 99.0 [78.0 to 126] | 39.0 [31.4 to 48.5]
  Serotype 2; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 2; Post-Injection 3 | 174 [139 to 218] | 157 [129 to 192]
  Serotype 3; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 3; Post-Injection 2 | 118 [101 to 139] | 37.9 [30.8 to 46.8]
  Serotype 3; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 3; Post-Injection 3 | 184 [158 to 214] | 160 [138 to 187]
  Serotype 4; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 4; Post-Injection 2 | 66.4 [51.8 to 85.1] | 24.0 [17.4 to 33.2]
  Serotype 4; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 4; Post-Injection 3 | 73.0 [60.0 to 88.7] | 72.2 [59.1 to 88.1]

12. Secondary Outcome: Percentage of FV-immune Participants With Antibody Titer >= 10 (1/Dil) Against Each Serotype With Parental Dengue Virus Strains After YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Neutralizing antibodies against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue PRNT assay. FV-immune participants at baseline were defined as those participants with >= 10 (1/dil) for at least 1 serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strain or for YF virus.
Time Frame: Pre-Injection 1 and 28 days Post-Injections 2 and 3
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 10 | 14
percentage of participants
  Serotype 1; Pre-Injection 1: number analyzed (Participants) | 10 | 13
  Serotype 1; Pre-Injection 1 | 10.0 | 0.0
  Serotype 1; Post-Injection 2 | 90.0 | 57.1
  Serotype 1; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 1; Post-Injection 3 | 100.0 | 100.0
  Serotype 2; Pre-Injection 1: number analyzed (Participants) | 10 | 12
  Serotype 2; Pre-Injection 1 | 20.0 | 0.0
  Serotype 2; Post-Injection 2 | 100.0 | 92.9
  Serotype 2; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 2; Post-Injection 3 | 100.0 | 100.0
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 8 | 13
  Serotype 3; Pre-Injection 1 | 12.5 | 30.8
  Serotype 3; Post-Injection 2 | 100.0 | 100.0
  Serotype 3; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 3; Post-Injection 3 | 100.0 | 100.0
  Serotype 4; Pre-Injection 1: number analyzed (Participants) | 10 | 13
  Serotype 4; Pre-Injection 1 | 0.0 | 7.7
  Serotype 4; Post-Injection 2 | 90.0 | 92.9
  Serotype 4; Post-Injection 3: number analyzed (Participants) | 9 | 13
  Serotype 4; Post-Injection 3 | 88.9 | 100.0

13. Secondary Outcome: Percentage of FV Non-immune (Naïve) Participants With Antibody Titer >= 10 (1/Dil) Against Each Serotype With the Parental Dengue Virus Strains After YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Neutralizing antibodies against each serotype (Serotype 1, 2, 3 and 4) with the parental dengue virus strains were assessed using a dengue PRNT assay. FV non-immune participants at baseline were defined as those participants with <10 (1/dil) for all serotypes (Serotype 1, 2, 3 and 4) with parental dengue virus strains and for YF virus.
Time Frame: Pre-Injection 1 and 28 days Post-Injections 2 and 3
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 94 | 90
Percentage of participants
  Serotype 1; Pre-Injection 1 | 0.0 | 0.0
  Serotype 1; Post-Injection 2 | 92.6 | 51.1
  Serotype 1; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 1; Post-Injection 3 | 100.0 | 96.5
  Serotype 2; Pre-Injection 1 | 0.0 | 0.0
  Serotype 2; Post-Injection 2 | 96.8 | 86.7
  Serotype 2; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 2; Post-Injection 3 | 100.0 | 100.0
  Serotype 3; Pre-Injection 1 | 0.0 | 0.0
  Serotype 3; Post-Injection 2 | 100.0 | 87.8
  Serotype 3; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 3; Post-Injection 3 | 100.0 | 100.0
  Serotype 4; Pre-Injection 1 | 0.0 | 0.0
  Serotype 4; Post-Injection 2 | 90.4 | 63.3
  Serotype 4; Post-Injection 3: number analyzed (Participants) | 93 | 86
  Serotype 4; Post-Injection 3 | 97.8 | 97.7

14. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site and Systemic Reactions Following Any and Each Injection With YF Vaccine (Stamaril®) Concomitantly With Either CYD Dengue Vaccine or a Placebo
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost and Irritability. Grade 3 Solicited injection site reactions: Tenderness: cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling: >=50 millimeter (mm). Grade 3 Solicited systemic reactions: Fever: >39.5°celsius; Vomiting: >= episodes per 24 hours or requiring parenteral hydration; Crying abnormal: >3 hours; Drowsiness: sleeping most of the time or difficult to wake up; Appetite lost: refuses >=3 feeds/meals or refuses most feeds/meals; Irritability: inconsolable. Solicited Injection site reaction were reported separately for Stamaril®, CYD and placebo vaccine.
Time Frame: Day 0 up to 14 days post any Inj., Post Inj. 1, Post Inj. 2 and Post Inj. 3
Population: Analysis was performed on Safety analysis set. Here, 'number analyzed' = participants with available data for each specified category. "0" in "number analyzed" field= none of the participants were evaluable since participants did not received CYD dengue vaccine as Injection 1 (Placebo group) or Placebo at any time point (CYD dengue vaccine group).
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 394 | 393
Percentage of participants
  Inj. site Tenderness for Stamaril®; Post-Any Inj.: number analyzed (Participants) | 386 | 386
  Inj. site Tenderness for Stamaril®; Post-Any Inj. | 25.4 | 17.6
  Grd 3 Inj. site Tenderness, Stamaril®;Post-Any Inj: number analyzed (Participants) | 386 | 386
  Grd 3 Inj. site Tenderness, Stamaril®;Post-Any Inj | 0.3 | 0.3
  Inj. site Tenderness for CYD dengue;Post-Any Inj.: number analyzed (Participants) | 386 | 363
  Inj. site Tenderness for CYD dengue;Post-Any Inj. | 36.5 | 28.9
  Grd 3 Inj site Tenderness, CYDdengue;Post-Any Inj: number analyzed (Participants) | 386 | 363
  Grd 3 Inj site Tenderness, CYDdengue;Post-Any Inj | 0.3 | 0.0
  Inj. site Tenderness for placebo; Post-Any Inj.: number analyzed (Participants) | 0 | 386
  Inj. site Tenderness for placebo; Post-Any Inj. |  | 19.7
  Grd 3 Inj. site Tenderness, placebo;Post-Any Inj.: number analyzed (Participants) | 0 | 386
  Grd 3 Inj. site Tenderness, placebo;Post-Any Inj. |  | 0.3
  Inj. site Erythema for Stamaril®; Post-Any Inj.: number analyzed (Participants) | 386 | 386
  Inj. site Erythema for Stamaril®; Post-Any Inj. | 8.3 | 9.8
  Grd 3 Inj. site Erythema, Stamaril®;Post-Any Inj.: number analyzed (Participants) | 386 | 386
  Grd 3 Inj. site Erythema, Stamaril®;Post-Any Inj. | 0.0 | 0.0
  Inj. site Erythema for CYD dengue;Post-Any Inj.: number analyzed (Participants) | 386 | 363
  Inj. site Erythema for CYD dengue;Post-Any Inj. | 12.7 | 8.8
  Grd 3 Inj. site Erythema, CYD dengue;Post-Any Inj: number analyzed (Participants) | 386 | 363
  Grd 3 Inj. site Erythema, CYD dengue;Post-Any Inj | 0.0 | 0.0
  Inj. site Erythema for placebo; Post-Any Inj.: number analyzed (Participants) | 0 | 386
  Inj. site Erythema for placebo; Post-Any Inj. |  | 10.9
  Grd 3 Inj. site Erythema for placebo; Post-Any Inj: number analyzed (Participants) | 0 | 386
  Grd 3 Inj. site Erythema for placebo; Post-Any Inj |  | 0.0
  Inj. site Swelling for Stamaril®; Post-Any Inj.: number analyzed (Participants) | 386 | 386
  Inj. site Swelling for Stamaril®; Post-Any Inj. | 4.7 | 4.4
  Grd 3 Inj. site Swelling, Stamaril®; Post-Any Inj.: number analyzed (Participants) | 386 | 386
  Grd 3 Inj. site Swelling, Stamaril®; Post-Any Inj. | 0.0 | 0.0
  Inj. site Swelling for CYD dengue; Post-Any Inj.: number analyzed (Participants) | 386 | 363
  Inj. site Swelling for CYD dengue; Post-Any Inj. | 7.5 | 6.1
  Grd 3 Inj. site Swelling, CYD dengue; Post-Any Inj: number analyzed (Participants) | 386 | 363
  Grd 3 Inj. site Swelling, CYD dengue; Post-Any Inj | 0.0 | 0.0
  Inj. site Swelling for placebo; Post-Any inj.: number analyzed (Participants) | 0 | 386
  Inj. site Swelling for placebo; Post-Any inj. |  | 4.9
  Grd 3 Inj. site Swelling for placebo; Post-Any Inj: number analyzed (Participants) | 0 | 386
  Grd 3 Inj. site Swelling for placebo; Post-Any Inj |  | 0.0
  Inj. site Tenderness for Stamaril®; Post-Inj. 1: number analyzed (Participants) | 386 | 386
  Inj. site Tenderness for Stamaril®; Post-Inj. 1 | 25.4 | 17.6
  Grd 3 Inj. site Tenderness, Stamaril®; Post-Inj. 1: number analyzed (Participants) | 386 | 386
  Grd 3 Inj. site Tenderness, Stamaril®; Post-Inj. 1 | 0.3 | 0.3
  Inj. site Tenderness for CYD dengue; Post-Inj. 1: number analyzed (Participants) | 386 | 0
  Inj. site Tenderness for CYD dengue; Post-Inj. 1 | 24.9 |
  Grd 3 Inj. site Tenderness, CYD dengue; Post-Inj 1: number analyzed (Participants) | 386 | 0
  Grd 3 Inj. site Tenderness, CYD dengue; Post-Inj 1 | 0.0 |
  Inj. site Tenderness for placebo; Post-Inj. 1: number analyzed (Participants) | 0 | 386
  Inj. site Tenderness for placebo; Post-Inj. 1 |  | 19.7
  Grd 3 Inj. site Tenderness, placebo; Post-Inj. 1: number analyzed (Participants) | 0 | 386
  Grd 3 Inj. site Tenderness, placebo; Post-Inj. 1 |  | 0.3
  Inj. site Erythema for Stamaril®; Post-Inj. 1: number analyzed (Participants) | 386 | 386
  Inj. site Erythema for Stamaril®; Post-Inj. 1 | 8.3 | 9.8
  Grd 3 Inj.site Erythema for Stamaril®; Post-Inj. 1: number analyzed (Participants) | 386 | 386
  Grd 3 Inj.site Erythema for Stamaril®; Post-Inj. 1 | 0.0 | 0.0
  Inj. site Erythema for CYD dengue; Post-Inj. 1: number analyzed (Participants) | 386 | 0
  Inj. site Erythema for CYD dengue; Post-Inj. 1 | 8.8 |
  Grd 3 Inj. site Erythema, CYD dengue; Post-Inj. 1: number analyzed (Participants) | 386 | 0
  Grd 3 Inj. site Erythema, CYD dengue; Post-Inj. 1 | 0.0 |
  Inj. site Erythema for placebo; Post-Inj. 1: number analyzed (Participants) | 0 | 386
  Inj. site Erythema for placebo; Post-Inj. 1 |  | 10.9
  Grd 3 Inj. site Erythema for placebo; Post-Inj. 1: number analyzed (Participants) | 0 | 386
  Grd 3 Inj. site Erythema for placebo; Post-Inj. 1 |  | 0.0
  Inj. site Swelling for Stamaril®; Post-Inj. 1: number analyzed (Participants) | 386 | 386
  Inj. site Swelling for Stamaril®; Post-Inj. 1 | 4.7 | 4.4
  Grd 3 Inj.site Swelling for Stamaril®; Post-Inj. 1: number analyzed (Participants) | 386 | 386
  Grd 3 Inj.site Swelling for Stamaril®; Post-Inj. 1 | 0.0 | 0.0
  Inj. site Swelling for CYD dengue; Post-Inj. 1: number analyzed (Participants) | 386 | 0
  Inj. site Swelling for CYD dengue; Post-Inj. 1 | 4.7 |
  Grd 3 Inj. site Swelling, CYD dengue; Post-Inj. 1: number analyzed (Participants) | 386 | 0
  Grd 3 Inj. site Swelling, CYD dengue; Post-Inj. 1 | 0.0 |
  Inj. site Swelling for placebo; Post-Inj. 1: number analyzed (Participants) | 0 | 386
  Inj. site Swelling for placebo; Post-Inj. 1 |  | 4.9
  Grd 3 Inj. site Swelling for placebo; Post-Inj. 1: number analyzed (Participants) | 0 | 386
  Grd 3 Inj. site Swelling for placebo; Post-Inj. 1 |  | 0.0
  Inj. site Tenderness for CYD dengue; Post-Inj. 2: number analyzed (Participants) | 371 | 363
  Inj. site Tenderness for CYD dengue; Post-Inj. 2 | 17.0 | 20.4
  Grd 3 Inj. site Tenderness, CYD dengue; Post-Inj 2: number analyzed (Participants) | 371 | 363
  Grd 3 Inj. site Tenderness, CYD dengue; Post-Inj 2 | 0.0 | 0.0
  Inj. site Erythema for CYD dengue; Post-Inj. 2: number analyzed (Participants) | 371 | 363
  Inj. site Erythema for CYD dengue; Post-Inj. 2 | 5.1 | 8.0
  Grd 3 Inj. site Erythema, CYD dengue; Post-Inj. 2: number analyzed (Participants) | 371 | 363
  Grd 3 Inj. site Erythema, CYD dengue; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Swelling for CYD dengue; Post-Inj. 2: number analyzed (Participants) | 371 | 363
  Inj. site Swelling for CYD dengue; Post-Inj. 2 | 2.7 | 4.7
  Grd 3 Inj. site Swelling, CYD dengue; Post-Inj. 2: number analyzed (Participants) | 371 | 363
  Grd 3 Inj. site Swelling, CYD dengue; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Tenderness for CYD dengue; Post-Inj. 3: number analyzed (Participants) | 364 | 355
  Inj. site Tenderness for CYD dengue; Post-Inj. 3 | 14.6 | 16.3
  Grd 3 Inj. site Tenderness, CYD dengue; Post-Inj 3: number analyzed (Participants) | 364 | 355
  Grd 3 Inj. site Tenderness, CYD dengue; Post-Inj 3 | 0.3 | 0.0
  Inj. site Erythema for CYD dengue; Post-Inj. 3: number analyzed (Participants) | 364 | 355
  Inj. site Erythema for CYD dengue; Post-Inj. 3 | 3.6 | 4.2
  Grd 3 Inj. site Erythema, CYD dengue; Post-Inj. 3: number analyzed (Participants) | 364 | 355
  Grd 3 Inj. site Erythema, CYD dengue; Post-Inj. 3 | 0.0 | 0.0
  Inj. site Swelling for CYD dengue; Post-Inj. 3: number analyzed (Participants) | 364 | 355
  Inj. site Swelling for CYD dengue; Post-Inj. 3 | 1.6 | 2.8
  Grd 3 Inj. site Swelling, CYD dengue; Post-Inj. 3: number analyzed (Participants) | 364 | 355
  Grd 3 Inj. site Swelling, CYD dengue; Post-Inj. 3 | 0.0 | 0.0
  Fever; Post-Any Injection: number analyzed (Participants) | 385 | 385
  Fever; Post-Any Injection | 48.1 | 40.3
  Grade 3 Fever; Post-Any Injection: number analyzed (Participants) | 385 | 385
  Grade 3 Fever; Post-Any Injection | 1.3 | 0.8
  Vomiting; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Vomiting; Post-Any Injection | 30.6 | 27.2
  Grade 3 Vomiting; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Grade 3 Vomiting; Post-Any Injection | 1.3 | 2.1
  Crying abnormal; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Crying abnormal; Post-Any Injection | 47.2 | 44.0
  Grade 3 Crying abnormal; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Grade 3 Crying abnormal; Post-Any Injection | 0.5 | 1.3
  Drowsiness; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Drowsiness; Post-Any Injection | 36.3 | 33.9
  Grade 3 Drowsiness; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Grade 3 Drowsiness; Post-Any Injection | 0.5 | 0.0
  Appetite lost; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Appetite lost; Post-Any Injection | 54.7 | 50.0
  Grade 3 Appetite lost; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Grade 3 Appetite lost; Post-Any Injection | 4.7 | 3.6
  Irritability; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Irritability; Post-Any Injection | 46.4 | 46.4
  Grade 3 Irritability; Post-Any Injection: number analyzed (Participants) | 386 | 386
  Grade 3 Irritability; Post-Any Injection | 1.6 | 1.6
  Fever; Post-Injection 1: number analyzed (Participants) | 378 | 375
  Fever; Post-Injection 1 | 26.7 | 16.5
  Grade 3 Fever; Post-Injection 1: number analyzed (Participants) | 378 | 375
  Grade 3 Fever; Post-Injection 1 | 1.1 | 0.3
  Vomiting; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Vomiting; Post-Injection 1 | 16.1 | 17.1
  Grade 3 Vomiting; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Grade 3 Vomiting; Post-Injection 1 | 0.5 | 1.0
  Crying abnormal; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Crying abnormal; Post-Injection 1 | 32.9 | 32.1
  Grade 3 Crying abnormal; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Grade 3 Crying abnormal; Post-Injection 1 | 0.5 | 1.3
  Drowsiness; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Drowsiness; Post-Injection 1 | 24.4 | 22.0
  Grade 3 Drowsiness; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Grade 3 Drowsiness; Post-Injection 1 | 0.5 | 0.0
  Appetite lost; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Appetite lost; Post-Injection 1 | 39.6 | 33.7
  Grade 3 Appetite lost; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Grade 3 Appetite lost; Post-Injection 1 | 4.4 | 3.1
  Irritability; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Irritability; Post-Injection 1 | 38.6 | 34.7
  Grade 3 Irritability; Post-Injection 1: number analyzed (Participants) | 386 | 386
  Grade 3 Irritability; Post-Injection 1 | 1.6 | 1.3
  Fever; Post-Injection 2: number analyzed (Participants) | 363 | 352
  Fever; Post-Injection 2 | 21.2 | 22.2
  Grade 3 Fever; Post-Injection 2: number analyzed (Participants) | 363 | 352
  Grade 3 Fever; Post-Injection 2 | 0.0 | 0.3
  Vomiting; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Vomiting; Post-Injection 2 | 12.4 | 8.8
  Grade 3 Vomiting; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Grade 3 Vomiting; Post-Injection 2 | 0.5 | 0.6
  Crying abnormal; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Crying abnormal; Post-Injection 2 | 19.7 | 21.8
  Grade 3 Crying abnormal; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Grade 3 Crying abnormal; Post-Injection 2 | 0.0 | 0.0
  Drowsiness; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Drowsiness; Post-Injection 2 | 12.7 | 16.5
  Grade 3 Drowsiness; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Grade 3 Drowsiness; Post-Injection 2 | 0.0 | 0.0
  Appetite lost; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Appetite lost; Post-Injection 2 | 27.0 | 23.1
  Grade 3 Appetite lost; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Grade 3 Appetite lost; Post-Injection 2 | 0.3 | 0.3
  Irritability; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Irritability; Post-Injection 2 | 17.3 | 22.3
  Grade 3 Irritability; Post-Injection 2: number analyzed (Participants) | 371 | 363
  Grade 3 Irritability; Post-Injection 2 | 0.0 | 0.0
  Fever; Post-Injection 3: number analyzed (Participants) | 344 | 332
  Fever; Post-Injection 3 | 20.3 | 17.8
  Grade 3 Fever; Post-Injection 3: number analyzed (Participants) | 344 | 332
  Grade 3 Fever; Post-Injection 3 | 0.3 | 0.3
  Vomiting; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Vomiting; Post-Injection 3 | 7.4 | 7.3
  Grade 3 Vomiting; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Grade 3 Vomiting; Post-Injection 3 | 0.3 | 0.6
  Crying abnormal; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Crying abnormal; Post-Injection 3 | 15.1 | 14.6
  Grade 3 Crying abnormal; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Grade 3 Crying abnormal; Post-Injection 3 | 0.0 | 0.0
  Drowsiness; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Drowsiness; Post-Injection 3 | 11.3 | 10.7
  Grade 3 Drowsiness; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Grade 3 Drowsiness; Post-Injection 3 | 0.0 | 0.0
  Appetite lost; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Appetite lost; Post-Injection 3 | 19.8 | 18.6
  Grade 3 Appetite lost; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Grade 3 Appetite lost; Post-Injection 3 | 0.0 | 0.3
  Irritability; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Irritability; Post-Injection 3 | 14.3 | 16.1
  Grade 3 Irritability; Post-Injection 3: number analyzed (Participants) | 364 | 355
  Grade 3 Irritability; Post-Injection 3 | 0.0 | 0.3

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from Day 0 (post-vaccination) of Month 0 up to 6 months post-Injection 3 (up to 573 days).
Description: A solicited reaction (SR) was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Safety analysis set.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/394 | 1/393
Serious Adverse Events (participants affected / at risk) | 35/394 | 38/393
Other Adverse Events (participants affected / at risk) | 211/394 | 193/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=394) | Placebo Group (N=393)
Accidental exposure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 6 (7) | 4 (4)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 12 (16) | 11 (11)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=394) | Placebo Group (N=393)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 18 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 22 (24)
Drowsiness; Post-Any Injection (Nervous system disorders) | 140/386 (182) | 131/386 (183)
Injection site Tenderness for Stamaril® vaccine; Post-Any Injection (General disorders) | 98/386 (98) | 68/386 (68)
Injection site Tenderness for CYD dengue vaccine; Post-Any Injection (General disorders) | 141/386 (212) | 105/363 (132)
Injection site Tenderness for placebo; Post-Any Injection (General disorders) | 0 (0) | 76/386 (76)
Injection site Erythema for Stamaril® vaccine; Post-Any Injection (General disorders) | 32/386 (32) | 38/386 (38)
Injection site Erythema for CYD dengue vaccine; Post-Any Injection (General disorders) | 49/386 (66) | 32/363 (44)
Injection site Erythema for placebo; Post-Any Injection (General disorders) | 0 (0) | 42 (42)
Injection site Swelling for CYD dengue vaccine; Post-Any Injection (General disorders) | 29/386 (34) | 22/363 (27)
Fever; Post-Any Injection (General disorders) | 185/385 (248) | 155/385 (199)
Crying abnormal; Post-Any injection (Psychiatric disorders) | 182 (255) | 170 (255)
Irritability; Post-Any injection (Psychiatric disorders) | 179 (265) | 179 (272)
Diarrhoea (Gastrointestinal disorders) | 61 (73) | 59 (71)
Vomiting; Post-Any injection (Gastrointestinal disorders) | 118/386 (135) | 105/386 (124)
Appetite lost; Post-Any injection (Metabolism and nutrition disorders) | 211 (325) | 193 (280)
Gastroenteritis (Infections and infestations) | 44 (46) | 43 (49)
Nasopharyngitis (Infections and infestations) | 118 (140) | 120 (140)
Pharyngitis (Infections and infestations) | 73 (90) | 52 (65)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.